CLINICAL TRIAL: NCT00212927
Title: The Association of Provider Continuity and Information Continuity With Patient Outcomes After Discharge From Hospital
Brief Title: Continuity of Care and Outcomes After Discharge From Hospital
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Other Study IDs: carl001
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2007-07

CONDITIONS: Patient Safety

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
1. INTRODUCTION: Continuity of care (COC) occurs when separate elements of patient care are connected. COC is made up primarily of Continuity of Provider (COP) and Continuity of Information (COI). Many authorities believe that COC is essential to high-quality care. Previous studies have shown poor COC in varied populations. Many studies have shown that increased COC has been associated with improved intermediate outcomes. However, no study has definitively determined whether COC or either of its components is associated with important outcomes. The Ontario-Outcomes After the Hospitalization (Ontario-OAtH) study will enroll 5900 adults who are discharged to the community from medical and surgical services from 13 teaching and community hospitals in 5 regions across Ontario. Patients will be followed for 6 months to record details about all interactions with the health care system. This information will give us a detailed measure of both provider and information continuity for all patients over time. The Ontario-OAtH study will have the power to precisely determine whether COC is associated with time to urgent readmission or death after hospital discharge. Since COC is potentially modifiable, the Ontario-OAtH study will give us essential information required for designing interventions to improve outcomes for patients after they are discharged from hospital.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* discharged to the community from medical and surgical services

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5900 (Estimated)
Dates: Start 2002-10; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Van Walraven, MD, Principal Investigator — OHRI
Locations (1):
- Ottawa Health Research Institute, Ottawa, Ontario, Canada